CLINICAL TRIAL: NCT02151370
Title: Ascites Control Treating Ovarian Cancer With Bevacizumab: "ACT-OB"
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28428
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will collect data about safety in female patients with advanced ovarian epithelial cancer with measurable residual disease after surger y. The treating physician has decided to treat the patients with Avastin (bevaci zumab) in combination with chemotherapy followed by Avastin monotherapy accordin g to the local label. Data will be collected for 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years of age
* Histologically confirmed Advanced Epithelial Ovarian Cancer
* Confirmed ascites prior to surgery
* Residual disease after surgery
* Patients are chemotherapy naïve or have received only one prior line of treatment for their disease
* International Federation of Gynecology and Obstetrics (FIGO) stage IIIb or IV disease
* Eastern Cooperative Oncology Group (ECOG) performance status <=2
* Patients must meet treatment eligibility requirements according to treating physician and Summary of Product Characteristics (SmPC) criteria for Avastin plus chemotherapy.

Exclusion Criteria:

* Pregnancy or lactation
* Low grade tumors, since this does not necessarily requires systemic treatment. Complete surgical resection
* Uncontrollable hypertension
* Unexplained bleeding
* Known hypersensitivity to any components of bevacizumab
* All contraindications specified in the respective Summary of Product Characteristics (SmPC) and/or local labelling of Avastin and the corresponding chemotherapy must be adhered to by the physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with Advanced FIGO Stage (IIIb to IV) Ovarian Epithelial Cancer with measurable residual disease after surgery
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who require paracenthesis during treatment with Avastin | 72 weeks
The amount of ascitic fluid extracted during treatment with Avastin | 72 weeks

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 72 weeks
To evaluate Eastern Cooperative Oncology Group (ECOG) performance status before and after start of therapy | 72 weeks
To determine regional epidemiologic data for the studied population | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- San Salvador, El Salvador